CLINICAL TRIAL: NCT04737382
Title: Osimertinib Resistance Analysis in Patients With EGFR Mutation Positive Non-small-cell Lung Carcinoma That Have Progressed on Osimertinib Treatment'
Brief Title: Osimertinib Resistance in Patients With Non-small-cell Lung Carcinoma That Have Progressed.
Acronym: OSIRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M18OSI
Record Dates: First submitted 2019-10-24; First posted 2021-02-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Non-small-cell Lung Carcinoma
Keywords: Osimertinib; EGFR positive NSCLC; Resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy and blood (Other): A histological core biopsy of a tumor lesion and a blood sample for ctDNA analysis will be collected
  Interventions: Diagnostic Test: biopsy; Diagnostic Test: ctDAN analysis

INTERVENTIONS:
Diagnostic Test: biopsy — The formalin fixed material will be processed for molecular analysis in a clinically validated diagnostic pipeline according to ISO 15189 or other acceptable standard
Diagnostic Test: ctDAN analysis — ctDNA analysis will be performed using the AVENIO ctDNA targeted kit according to the guidelines from the manufacturer with respect to isolation, library preparation and bioinformatics analysis.

SUMMARY:
Initially, patients with EGFR mutation positive NSCLC respond well to osimertinib, a third generation EGFR tyrosine kinase inhibitor (TKI), but eventually progress. Upon progression multiple resistance mechanisms have been described and new therapeutic strategies are being developed to target these resistance mechanisms. Thorough and complete osimertinib resistance analysis enables optimal treatment decision making and might identify new targets for molecular treatment, thereby potentially improving patient outcome.

DETAILED DESCRIPTION:
Initially, patients with EGFR mutation positive NSCLC respond well to osimertinib, a third generation EGFR tyrosine kinase inhibitor (TKI), but eventually progress. Upon progression, three main resistance mechanisms can be found (1, 2): 1) alteration of the drug target by secondary or tertiary EGFR mutations (e.g. C797S mutation in the EGFR kinase domain), 2) alteration of downstream signal transduction proteins (e.g. KRAS mutation / amplification) and 3) bypass track resistance like MET or HER2 amplification. A fourth, less frequent, mechanism involves morphological alterations: dedifferentiation by epidermal-mesenchymal transition (EMT) or change to small-cell-lung carcinoma (SCLC), including RB1 loss.

New therapeutic strategies are being developed to target these resistance mechanisms and reports have been published about successful treatment of HER2 and MET amplification. Drugs targeting the C797S mutation are entering the clinic.

Next Generation Sequence (NGS) technology rapidly evolves and it is now feasible to analyse broad panels of genetic alterations in tumor tissue as well as in circulating tumor DNA (ctDNA).

ctDNA based T790M detection is a valid method to test for resistance to first or second generation EGFR TKI's and the ctDNA based technique is increasingly being used for patients with progression on the third generation EGFR TKI osimertinib. Actually, the distribution of osimertinib resistance mechanisms, as known to date, largely comes from ctDNA based datasets, because biopsy based analyses are scarce. Due to impaired sensitivity of ctDNA based analyses when compared to tissue based analysis, especially for copy number variations, these reports might be misleading and lead to suboptimal treatment. Early reports of tumor samples obtained after progression on first / second generation EGFR TKI's have shown that ctDNA and tumor based drug resistance analyses can be concordant or disconcordant and that the tests should be regarded as complimentary [Oxnard et al].

Sensitivity and specificity of ctDNA and biopsy based drug resistance analysis after osimertinib treatment and how these tests behave within individual patients are unknown.

Thorough and complete osimertinib resistance analysis enables optimal treatment decision making and might identify new targets for molecular treatment, thereby potentially improving patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic NSCLC, characterized by a sensitizing EGFR mutation.

  2. Progressive disease, as assessed by the treating physician during osimertinib monotherapy.

  3. Eligible for subsequent treatment. 4. Willing to undergo a histological biopsy and withdrawal of a blood sample for ctDNA analysis.

  5. Technically possible to take a histological biopsy.

Exclusion Criteria:

- 1. Osimertinib discontinuation before blood draw and / or histological tumor biopsy.

2. Initiation of a new line of anticancer therapy before blood draw and / or histological tumor biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2024-08-22 (Estimated); Study Completion 2024-08-22 (Estimated)

PRIMARY OUTCOMES:
EGFR TKI resistance analysis on tumor biopsies and ctDNA | Trough study completion, an average of 2 years
  Complete osimertinib resistance analysis in tissue and plasma for all patients in the Netherlands that progress on osimertinib treatment
Recommendation for subsequent treatment | Trough study completion, an average of 2 years
  Evaluation of these results in an MTB meeting and recommendations for subsequent treatment.

SECONDARY OUTCOMES:
Evaluate recommended and actually treatment | Trough study completion, an average of 2 years
  Number of patients with concordant recommended and actually provided subsequent treatment.
Evaluate plasma and tumor tissue | Trough study completion, an average of 2 years
  Number of patients with concordance in osimertinib resistance in plasma using ctDNA and in tumor tissue.
Evaluate success rate | Trough study completion, an average of 2 years
  To evaluate the success rate of molecular profiling on tumor tissue and ctDNA (test successfully performed or not).

CONTACTS AND LOCATIONS:
Overall Officials: J de Langen, MD, PhD, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek
Locations (6):
- Netherlands (6):
  - The Netherlands Cancer Institute-Antoni van Leeuwenhoek, Amsterdam, North Holland
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus MC, Universitair Medisch Centrum Rotterdam, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Wel JWT, Ernst SM, Jebbink M, van den Broek D, Badrising SK, Steinbusch LC, Ruiter G, Theelen WSME, van Veggel BAMH, Smit J, Dingemans AM, Paats MS, Dubbink HJ, Hashemi SMS, Radonic T, Cohen D, van der Wekken AJ, Ter Elst A, Timens W, Hendriks LE, Speel EJM, Disselhorst MMJ, Welling A, van der Meer F, Bosch LJW, Monkhorst K, Boelens MC, Smit EF, de Langen AJ. Determining the optimal approach to identify osimertinib resistance; the first line osimertinib cohort of the OSIRIS study. Lung Cancer. 2025 Nov;209:108783. doi: 10.1016/j.lungcan.2025.108783. Epub 2025 Sep 28. PMID 41039677